CLINICAL TRIAL: NCT04118478
Title: Effects of Multicomponent Exercise Program With Progressive Phases on Functional Capacity, Fitness, Quality of Life, Dual-Task and Physiological Variables in Older Adults: Randomized Controlled Trial Protocol
Brief Title: Effect of a Multi-component Training Program With Progressive Phases on the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Emilio Eduardo Jofre Saldia, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EJofre
Record Dates: First submitted 2019-09-30; First posted 2019-10-08 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: ELDERLY PEOPLE
Keywords: fitness; program training; exercise; health; physical condition; qualilty of Life; Functional capacity; physiological status; physical activity; elderly
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A study protocol of a randomized controlled clinical trial with blinded examiners is presented.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The investigator performing the randomization will be blinded and will not participate in the recruitment process. Participants and group assignment will be blinded to investigators and technicians performing statistical analysis. Participants will be explicitly informed of their assigned group, without the possibility of modification throughout the program. The evaluation team will be made up of five researchers and technicians, two will apply the different phases of the program, one will randomly assign the participants and two others will oversee the statistical analysis. All the analysis of the results will be gathered by the same researcher. The researcher will neither know which group the participant belongs to, nor the main design of the study or the foreseen changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-component phased training program (Experimental): The intervention of the program consists of conducting a multi-component training in a neighborhood unit.
  The intervention will consist of the realization of a multi-component program in a training center adapted for the elderly. The duration of the program will be 27 weeks with a frequency of two weekly sessions and an intervention duration of 45 to 60 minutes
  Interventions: Behavioral: multi-component phased training program
- CONTROL (No Intervention): Older people assigned to the GC do not do any training programming. Only attend the measurement dates.

INTERVENTIONS:
Behavioral: multi-component phased training program — The experimental group will develop a program that consists of three progressive phases with the predominance of one physical quality over the others. The first phase will have as its main objective to develop strength, through exercises with overload and in turn, it will be subdivided into 3 blocks of 3 weeks each: Neuromuscular adaptation, muscular power, muscular resistance. The second phase will have as its main objective to develop cardiorespiratory capacity through intermittent gait training and, in turn, will be subdivided into 3 blocks of 3 weeks each: Static gait, dynamic gait and dynamic gait with changes of direction. The last phase will have as its main objective to develop balance and flexibility, by strengthening the stabilizing muscles and range of motion. In turn, this phase will be subdivided into 3 blocks of 3 weeks each: Balance / static flexibility, balance / dynamic flexibility and balance / flexibility with a double task.
  Arms: Multi-component phased training program

SUMMARY:
The increase in life expectancy worldwide, added to the decrease in birth rates, has resulted in an increase in the aging population. In the case of Chile, 11.4% of its inhabitants are older adults and specifically, in the Til-Til commune, 14.65% of the total population is over 60 years of age, directly affecting the neuromuscular system and mainly cardiorespiratory. Therefore, the older person lives longer, but with a lower quality of life. Physical exercise appears as a non-pharmacological alternative to improve the quality of life, physical and cognitive functions. The "multi-component training" consists of a program that combines strength, resistance, balance and gait training, and is the one that presents the greatest improvements in the functional capacity of the elderly person.

The objective of the present investigation is to relate the effects of a multi-component training schedule by phases on the quality of life, functional capacity and physiological parameters in a group of people over 60 to 80 years of age in the commune of Til-Til.

DETAILED DESCRIPTION:
The intervention consists of carrying out a 27-week multi-component training program divided into 3 phases of 9 weeks each, where the physical qualities will be progressively worked together twice a week. However, in each phase the development of one physical quality will predominate over the others. Each session will be supervised by two experienced physical educators in the area, they will also be trained two weeks prior to the intervention and supervised weekly by the principal investigator. The first phase will have as its main objective to develop strength, through exercises with overload and in turn, it will be subdivided into 3 blocks of 3 weeks each: Neuromuscular adaptation (block 1), muscular power (block 2), muscular resistance (block 3). Each session will last approximately 45 minutes at an intensity of 70-75% of one maximum repetition (1RM) and with an effort character from light to maximum. The session will consist of 10 minutes of mobility and muscle activation as a warm-up, 25 minutes of strength exercises and 10 minutes of stretching as a return to calm. The second phase will have as its main objective to develop cardiorespiratory capacity through intermittent gait training and, in turn, will be subdivided into 3 blocks of 3 weeks each: Static gait (block 1), dynamic gait (block 2) and dynamic gait with changes of direction (block 3). Each session will last approximately 50 minutes with an effort perception of 6-8. The session will consist of 10 minutes of mobility and muscular activation as a warm-up, 10 minutes of muscular power exercises, 20 minutes of cardiorespiratory endurance and 10 minutes of stretching as a return to calm. The last phase will have as its main objective to develop balance and flexibility, by strengthening the stabilizing muscles and range of motion. In turn, this phase will be subdivided into 3 blocks of 3 weeks each: Balance / static flexibility (block 1), balance / dynamic flexibility (block 2) and balance / flexibility with a double task (block 3). Each session will last approximately 60 minutes with a perception of effort of 6-8. The session will consist of 10 minutes of mobility and muscle activation as a warm-up, 10 minutes of power exercises, 10 minutes of cardiorespiratory endurance, 20 minutes of balance exercises and 10 minutes of stretching as a return to calm).

ELIGIBILITY:
The inclusion criteria are: a) being between 60 to 80 years old, b) being able to move with or without personal / technical assistance, c) able to communicate, d) autonomy to give consent or, otherwise, be assisted by a relative or legal representative. Exclusion criteria are any factors that exclude the performance of the physical training program or testing procedures as determined by the treating physician. These factors include, but are not limited to, the following: a) terminal disease, b) acute myocardial infarction in the past 3 months, c) unstable cardiovascular disease or other medical condition, d) fracture of the upper or lower extremity in the last 3 months, e) severe dementia, f) unwillingness to complete study requirements or to be randomized to the control or intervention group.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Assessment of the quality of life | Change from Baseline quality life at 2, 4 and at 6 month
  The quality of life will be assessed through the SF-36 health questionnaire, which represents a generic scale that provides a profile of the state of health and is applicable to both patients and the general population.
Heart rate variability | Change from Baseline Heart rate variability at 2, 4 and at 6 month
  The heart rate variability (CRV) corresponds to an indicator of the modulation exerted by the autonomic nervous system, which will be analyzed in the frequency and time domains and represents an adequate analysis of the variation from beat to beat, from a point of temporal view, expressing differences in the consecutive RR intervals of the QRS complexes of an electrocardiogram. The VRC will be registered using the HRV Expert Cardiomood® smartphone application, which is capable of recording the RR intervals for analysis of the VRC indexes with high level of reliability (R = 0.97) and the H7® POLAR model heart rate monitor capable of recording these intervals as reliably (r = 0.99) as an electrocardiogram (ECG) test
Spirometry, forced expiratory volume in one second (FEV1) | Change from Baseline Spirometry FEV1 at 2, 4 and at 6 month
  Spirometry is a fundamental test in functional respiratory evaluation, which is frequently used in clinical practice and in population studies, due to its good reproducibility, ease of measurement and its degree of correlation with the stage of the disease, functional condition , morbidity and mortality.
  Forced Espiratory Volume1, (FEV1): Amount of air that mobilizes in the first second of an expiration forced. It is a flow, not a volume (milliliters / 1 sg), so which can be expressed as ml / s or as a percentage in front of his theoretical figures. Its normal value is greater than 80% The device used to measure this pulmonary parameter will be the Manual Spirometer CMS-SP10® of small volume and easy application.
Spirometry, peak expiratory flow (PEF) | Change from Baseline Spirometry PEF at 2, 4 and at 6 month
  Spirometry is a fundamental test in functional respiratory evaluation, which is frequently used in clinical practice and in population studies, due to its good reproducibility, ease of measurement and its degree of correlation with the stage of the disease, functional condition , morbidity and mortality. Peak Espiratory Flow, (PEF): Maximum amount of air that can be exhaled by second in a forced expiration. It is the maximum peak of flow which is obtained (flow - volume curve), and is produced before having expelled 15% of the FVC. It is a marker especially useful in the diagnosis of asthma and in crises asthmatics, where predictive target value of gravity. It is measured in liters / sec, or as a percentage of the reference value.
  The device used to measure this pulmonary parameter will be the Manual Spirometer CMS-SP10® of small volume and easy application.
Resting Heart rate | Change from Baseline Resting Heart rate at 2, 4 and at 6 month
  The heart rate (HR) is determined by the balance between the sympathetic and parasympathetic systems, which responds to the body's needs at all times.
Resting blood pressure | Change from resting blood pressure at 2, 4 and at 6 month
  Blood pressure (BP) shows a progressive increase with age and it is observed that systolic blood pressure shows a continuous increase, while diastolic pressure begins to decline after the age of 50 in both sexes.
Short Physical Performance Battery (SPPB) | Change from Baseline SPPB at 2, 4 and at 6 month
  It is a battery widely used in research and covers a wide spectrum of functional levels. It has proven its validity, reproducibility and sensitivity to change in different American and European populations with good results. It is composed of three subtests: one of balance (balance with feet together, in semi-tandem and in tandem), another of leg thrust (getting up and sitting from a chair without armrests five times as quickly as possible) and a third, consisting of measuring the normal speed of walking along 4 and 6 meters. The score ranges between 0 and 12 points, and scores between 4 and 9 are suggestive of fragility.
Walking speed in 4 and 6 meters | Change from Baseline Walking speed in 4 and 6 meters at 2, 4 and at 6 month
  Evaluation method that has taken great relevance recently and is even advocated as the simplest and most valid way of evaluation in the elderly. For its measurement, the time it takes for the older person to travel a certain distance is calculated (in the case of the present investigation it will be in 4 and 6 meters), and then it is passed to meters / second. It is usually evaluated at a normal pace, although it can also be done at a fast pace.
Time Up and Go | Change from Baseline Time Up and Go at 2, 4 and at 6 month
  It is a tool to assess the mobility and function of the lower limb, which proves to be useful, practical, fast and simple, without requiring a special team or specific training by the evaluator. Measure the time in seconds the subject takes to get up from a chair, walk 3 meters, turn, walk back to normal pace and sit down. This test has a good correlation with the measures of balance, walking speed, functionality and cognition, especially with the executive functions, memory and processing speed.
Dynamometry | Change from Baseline Dynamometry at 2, 4 and at 6 month
  The use of the dynamometer allows to determine the maximum isometric force in different muscle groups. Among them, the measurement of the pressing force of the dominant hand is especially important, given that it is a simple and non-invasive marker of muscular strength of the upper extremities.
Walking While Talking (WWT) | Change from Baseline Walking While Talking at 2, 4 and at 6 month
  This test will evaluate the speed of travel under the condition of counting backwards (from number 20 backwards) while walking at a distance of 6 meters, which has been proposed as a better instrument for measuring the speed of travel, because to which adds conditions of stress, difficulty or distraction, which presents a greater sensitivity to detect early mobility problems or preclinical disability
Two minutes "Step test" | Change from Baseline Two minutes "Step test" at 2, 4 and at 6 month
  The test consists of performing the greatest number of steps marching in place for two minutes, each knee reaching an intermediate point between the patella and the anterior superior iliac spine. Although both knees must reach the correct height, only the number of times the right knee reaches the determined height is counted
Sit and reach test | Change from Baseline Sit and reach test at 2, 4 and at 6 month
  This test will measure the flexibility of the lower body, mainly the biceps femoris and the lower back. It is an adapted version of the Wells test that measures the flexibility of both legs simultaneously, to an alternative consisting of evaluating only one lower limb sitting in a chair.
Back scratch test | Change from Baseline Back scratch test at 2, 4 and at 6 month
  This test will assess the flexibility of the upper body, specifically the mobility of the shoulder joint and validly shows the expected reduction in shoulder flexibility in subjects aged 60 to 80 years.

SECONDARY OUTCOMES:
Motivation for the exercise | Change from Baseline Motivation for the exercise at 6 month
  The motivation for the physical exercise will be evaluated through the Questionnaire of the Regulation of the Conduct in the Exercise (BREQ-3), which is headed by the sentence "I do physical exercise ..." in 23 items: Four for intrinsic regulation , four for integrated regulation ("because it agrees with my way of life", "because I consider that physical exercise is part of me", "because I see physical exercise as a fundamental part of who I am", "because I consider that the physical exercise is in accordance with my values "), three for identified regulation, four for introjected regulation, four for external regulation and four for demotivation.
"Physical Activity Vital Sign" (PAVS) | Change from Baseline "Physical Activity Vital Sign" at 6 month
  The level of physical activity will be recorded through two questionnaire: "Vital Sign of Physical Activity" (SVAF). The SVAF was developed as a simple questionnaire for use in a clinical setting with the objective of assessing moderate to vigorous physical activity (AFMV) of the last week and of a typical (usual) week.
"Stanford Short Activity Survey" | Change from Baseline "Stanford Short Activity Survey" at 6 month
  "Stanford Short Activity Survey" was developed to classify the levels of physical activity at work and during leisure time. The study used five brief descriptions of physical activity profiles, which are named inactive at high levels of commitment to exercise. Respondents select one profile for work and another for free time.
Abdominal circumference | Change from Baseline Abdominal circumference at 2, 4 and at 6 month
  The measurement will be performed with a SECA S201® measuring tape with an accuracy of 0.1 cm. The tape will be located in the midpoint between the internal rib edge of the last rib intercepted with the anterior axillary line and the iliac crest and it will be verified that the person is not inspired or forced expiration, registering the waist circumference obtained in centimeters .
Electrical impedance | Change from Baseline Electrical impedance at 2, 4 and at 6 month
  It is a safe, fast, simple, non-invasive procedure and with a good correlation with more complex techniques. Studies have shown that electrical bioimpedance is a safe, reproducible and reliable method to assess body composition. The instrument to be used for research is the OMRON HBF-514® model.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Jofré-Saldía, MSc, Principal Investigator — UCAM; Gemma García, Phd, Study Director — UCAM; Alvaro Villalobos, Msc, Principal Investigator — University of Ibadan Teaching Hospital (UCH)
Locations (1):
- Universidad Catolica de murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ball TJ, Joy EA, Gren LH, Shaw JM. Concurrent Validity of a Self-Reported Physical Activity "Vital Sign" Questionnaire With Adult Primary Care Patients. Prev Chronic Dis. 2016 Feb 4;13:E16. doi: 10.5888/pcd13.150228. PMID 26851335
- [Background] Bouaziz W, Vogel T, Schmitt E, Kaltenbach G, Geny B, Lang PO. Health benefits of aerobic training programs in adults aged 70 and over: a systematic review. Arch Gerontol Geriatr. 2017 Mar-Apr;69:110-127. doi: 10.1016/j.archger.2016.10.012. Epub 2016 Oct 31. PMID 27912156
- [Background] Cabrero-Garcia J, Munoz-Mendoza CL, Cabanero-Martinez MJ, Gonzalez-Llopis L, Ramos-Pichardo JD, Reig-Ferrer A. [Short physical performance battery reference values for patients 70 years-old and over in primary health care]. Aten Primaria. 2012 Sep;44(9):540-8. doi: 10.1016/j.aprim.2012.02.007. Epub 2012 May 16. Spanish. PMID 22608368
- [Background] Cadore EL, Menger E, Teodoro JL, da Silva LXN, Boeno FP, Umpierre D, Botton CE, Ferrari R, Cunha GDS, Izquierdo M, Pinto RS. Functional and physiological adaptations following concurrent training using sets with and without concentric failure in elderly men: A randomized clinical trial. Exp Gerontol. 2018 Sep;110:182-190. doi: 10.1016/j.exger.2018.06.011. Epub 2018 Jun 13. PMID 29908345
- [Background] Chan WC, Yeung JW, Wong CS, Lam LC, Chung KF, Luk JK, Lee JS, Law AC. Efficacy of physical exercise in preventing falls in older adults with cognitive impairment: a systematic review and meta-analysis. J Am Med Dir Assoc. 2015 Feb;16(2):149-54. doi: 10.1016/j.jamda.2014.08.007. Epub 2014 Oct 7. PMID 25304179
- [Background] Coelho-Junior HJ, de Oliveira Goncalvez I, Sampaio RAC, Sewo Sampaio PY, Cadore EL, Izquierdo M, Marzetti E, Uchida MC. Periodized and non-periodized resistance training programs on body composition and physical function of older women. Exp Gerontol. 2019 Jul 1;121:10-18. doi: 10.1016/j.exger.2019.03.001. Epub 2019 Mar 9. PMID 30862526
- [Background] Fragala MS, Cadore EL, Dorgo S, Izquierdo M, Kraemer WJ, Peterson MD, Ryan ED. Resistance Training for Older Adults: Position Statement From the National Strength and Conditioning Association. J Strength Cond Res. 2019 Aug;33(8):2019-2052. doi: 10.1519/JSC.0000000000003230. PMID 31343601
- [Background] Gomez-Morales A, Miranda JMA, Pergola-Marconato AM, Mansano-Schlosser TC, Mendes FRP, Torres GV. [The influence of activities on the quality of life of the elderly: a systematic review]. Cien Saude Colet. 2019 Jan;24(1):189-202. doi: 10.1590/1413-81232018241.05452017. Spanish. PMID 30698253
- [Background] Guizelini PC, de Aguiar RA, Denadai BS, Caputo F, Greco CC. Effect of resistance training on muscle strength and rate of force development in healthy older adults: A systematic review and meta-analysis. Exp Gerontol. 2018 Feb;102:51-58. doi: 10.1016/j.exger.2017.11.020. Epub 2017 Nov 28. PMID 29196141
- [Background] Izquierdo M. [Multicomponent physical exercise program: Vivifrail]. Nutr Hosp. 2019 Jul 1;36(Spec No2):50-56. doi: 10.20960/nh.02680. Spanish. PMID 31189323
- [Background] Joseph RP, Keller C, Adams MA, Ainsworth BE. Validity of two brief physical activity questionnaires with accelerometers among African-American women. Prim Health Care Res Dev. 2016 May;17(3):265-76. doi: 10.1017/S1463423615000390. Epub 2015 Jul 16. PMID 26178779
- [Background] Kim BS, Kim JH, Park SH, Seo HS, Lee HS, Lee MM. Effect of a Respiratory Training Program Using Wind Instruments on Cardiopulmonary Function, Endurance, and Quality of Life of Elderly Women. Med Sci Monit. 2018 Jul 29;24:5271-5278. doi: 10.12659/MSM.909492. PMID 30056459
- [Background] Lu WC, Tzeng NS, Kao YC, Yeh CB, Kuo TB, Chang CC, Chang HA. Correlation between health-related quality of life in the physical domain and heart rate variability in asymptomatic adults. Health Qual Life Outcomes. 2016 Oct 21;14(1):149. doi: 10.1186/s12955-016-0555-y. PMID 27765048
- [Background] Marcos-Pardo PJ, Orquin-Castrillon FJ, Gea-Garcia GM, Menayo-Antunez R, Gonzalez-Galvez N, Vale RGS, Martinez-Rodriguez A. Effects of a moderate-to-high intensity resistance circuit training on fat mass, functional capacity, muscular strength, and quality of life in elderly: A randomized controlled trial. Sci Rep. 2019 May 24;9(1):7830. doi: 10.1038/s41598-019-44329-6. PMID 31127163
- [Background] Mendonca GV, Pezarat-Correia P, Vaz JR, Silva L, Almeida ID, Heffernan KS. Impact of Exercise Training on Physiological Measures of Physical Fitness in the Elderly. Curr Aging Sci. 2016;9(4):240-259. doi: 10.2174/1874609809666160426120600. PMID 27113585
- [Background] Millor N, Lecumberri P, Gomez M, Martinez A, Martinikorena J, Rodriguez-Manas L, Garcia-Garcia FJ, Izquierdo M. Gait Velocity and Chair Sit-Stand-Sit Performance Improves Current Frailty-Status Identification. IEEE Trans Neural Syst Rehabil Eng. 2017 Nov;25(11):2018-2025. doi: 10.1109/TNSRE.2017.2699124. Epub 2017 Apr 27. PMID 28463202
- [Background] Perez-Sousa MA, Venegas-Sanabria LC, Chavarro-Carvajal DA, Cano-Gutierrez CA, Izquierdo M, Correa-Bautista JE, Ramirez-Velez R. Gait speed as a mediator of the effect of sarcopenia on dependency in activities of daily living. J Cachexia Sarcopenia Muscle. 2019 Oct;10(5):1009-1015. doi: 10.1002/jcsm.12444. Epub 2019 May 8. PMID 31066999
- [Background] Raffin J, Barthelemy JC, Dupre C, Pichot V, Berger M, Feasson L, Busso T, Da Costa A, Colvez A, Montuy-Coquard C, Bouvier R, Bongue B, Roche F, Hupin D. Exercise Frequency Determines Heart Rate Variability Gains in Older People: A Meta-Analysis and Meta-Regression. Sports Med. 2019 May;49(5):719-729. doi: 10.1007/s40279-019-01097-7. PMID 30945205
- [Background] Ramirez-Campillo R, Alvarez C, Garcia-Hermoso A, Celis-Morales C, Ramirez-Velez R, Gentil P, Izquierdo M. Reply to the commentary on: High-speed resistance training in elderly women: Effects of cluster training sets on functional performance and quality of life. Exp Gerontol. 2019 Aug;123:34-35. doi: 10.1016/j.exger.2019.05.012. Epub 2019 May 25. No abstract available. PMID 31136812
- [Background] Ramirez-Velez R, Correa-Bautista JE, Garcia-Hermoso A, Cano CA, Izquierdo M. Reference values for handgrip strength and their association with intrinsic capacity domains among older adults. J Cachexia Sarcopenia Muscle. 2019 Apr;10(2):278-286. doi: 10.1002/jcsm.12373. Epub 2019 Mar 6. PMID 30843369
- [Background] Ramirez-Velez R, Izquierdo M. Editorial: Precision Physical Activity and Exercise Prescriptions for Disease Prevention: The Effect of Interindividual Variability Under Different Training Approaches. Front Physiol. 2019 May 24;10:646. doi: 10.3389/fphys.2019.00646. eCollection 2019. No abstract available. PMID 31178759
- [Background] Rodriguez-Manas L, Laosa O, Vellas B, Paolisso G, Topinkova E, Oliva-Moreno J, Bourdel-Marchasson I, Izquierdo M, Hood K, Zeyfang A, Gambassi G, Petrovic M, Hardman TC, Kelson MJ, Bautmans I, Abellan G, Barbieri M, Pena-Longobardo LM, Regueme SC, Calvani R, De Buyser S, Sinclair AJ; European MID-Frail Consortium. Effectiveness of a multimodal intervention in functionally impaired older people with type 2 diabetes mellitus. J Cachexia Sarcopenia Muscle. 2019 Aug;10(4):721-733. doi: 10.1002/jcsm.12432. Epub 2019 Apr 23. PMID 31016897
- [Background] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Casas-Herrero A, Ramirez-Velez R, Izquierdo M. Role of muscle power output as a mediator between gait variability and gait velocity in hospitalized older adults. Exp Gerontol. 2019 Sep;124:110631. doi: 10.1016/j.exger.2019.110631. Epub 2019 Jun 12. PMID 31201920
- [Background] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Casas-Herrero A, Izquierdo M. Role of physical exercise on cognitive function in healthy older adults: A systematic review of randomized clinical trials. Ageing Res Rev. 2017 Aug;37:117-134. doi: 10.1016/j.arr.2017.05.007. Epub 2017 Jun 3. PMID 28587957
- [Background] Tan JPH, Beilharz JE, Vollmer-Conna U, Cvejic E. Heart rate variability as a marker of healthy ageing. Int J Cardiol. 2019 Jan 15;275:101-103. doi: 10.1016/j.ijcard.2018.08.005. Epub 2018 Aug 3. PMID 30104034
- [Background] Taylor-Piliae RE, Fair JM, Haskell WL, Varady AN, Iribarren C, Hlatky MA, Go AS, Fortmann SP. Validation of the Stanford Brief Activity Survey: examining psychological factors and physical activity levels in older adults. J Phys Act Health. 2010 Jan;7(1):87-94. doi: 10.1123/jpah.7.1.87. PMID 20231759
- [Background] Teodoro JL, da Silva LXN, Fritsch CG, Baroni BM, Grazioli R, Boeno FP, Lopez P, Gentil P, Bottaro M, Pinto RS, Izquierdo M, Cadore EL. Concurrent training performed with and without repetitions to failure in older men: A randomized clinical trial. Scand J Med Sci Sports. 2019 Aug;29(8):1141-1152. doi: 10.1111/sms.13451. Epub 2019 May 22. PMID 31050048
- [Background] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162
- [Background] Ball TJ, Joy EA, Goh TL, Hannon JC, Gren LH, Shaw JM. Validity of two brief primary care physical activity questionnaires with accelerometry in clinic staff. Prim Health Care Res Dev. 2015 Jan;16(1):100-8. doi: 10.1017/S1463423613000479. Epub 2014 Jan 28. PMID 24472569
- [Derived] Jofre-Saldia E, Villalobos-Gorigoitia A, Gea-Garcia G. Effects of multicomponent exercise program with progressive phases on functional capacity, fitness, quality of life, dual-task and physiological variables in older adults: Randomized controlled trial protocol. Rev Esp Geriatr Gerontol. 2021 Sep-Oct;56(5):272-278. doi: 10.1016/j.regg.2021.04.006. Epub 2021 Jun 8. PMID 34112535